CLINICAL TRIAL: NCT02451280
Title: Unilateral vs. Bilateral Approaches to Hybrid Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-1621A3
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
Keywords: stroke rehabilitation; robot-assisted therapy; hybrid therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unilateral Hybrid Intervention Group (Experimental): Participants will receive 6 weeks of bilateral RT training using the BMT and UAT training in each session.
  Interventions: Procedure: Unilateral Hybrid Intervention
- Bilateral Hybrid Intervention Group (Experimental): Participants will receive 6 weeks of bilateral RT training using the BMT and BAT training in each session.
  Interventions: Procedure: Bilateral Hybrid Intervention
- Robot-Assisted Training Group (Experimental): Participants will receive 6 weeks of RT training using the BMT in each session.
  Interventions: Procedure: Robot-Assisted Training

INTERVENTIONS:
Procedure: Unilateral Hybrid Intervention — For the unilateral RT training, participants will practice with their affected arms following a unilateral training protocol of BMT for 45 minutes (Yang, et al., 2012). For the UAT training, participants will receive training of the affected UL in functional tasks with behavioral shaping for 45 minutes (Lin, Wu, et al., 2009).
  Arms: Unilateral Hybrid Intervention Group
Procedure: Bilateral Hybrid Intervention — For the bilateral RT training, patients will focus on training involving both arms using the BMT robot for 45 minutes. During the 45 minutes BAT training, participants will receive training in tasks focusing on bilateral symmetric or alternating movements of both ULs.
  Arms: Bilateral Hybrid Intervention Group
Procedure: Robot-Assisted Training — The RT intervention will be matched in duration and intensity with the hybrid interventions. Participants in the RT group will practice on the BMT with bilateral protocols for 90 minutes. The tasks will be tailored according to the level
  Arms: Robot-Assisted Training Group

SUMMARY:
The aim of the project is to compare the effects of unilateral hybrid therapy [unilateral robot-assisted therapy (RT)] + unilateral arm training (UAT)] and bilateral hybrid therapy [bilateral RT + bilateral arm training (BAT)] on motor function, daily function, mobility, life quality, and motor control strategy in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥3 months onset from a first-ever unilateral stroke;
2. minimal motor criteria to receive CIT (i.e., ≥10º wrist extension and ≥ 10º extension at the thumb and any two other digits);
3. an initial FMA-UE score of 10 to 56, indicating mild to moderate and moderate to severe upper extremity motor impairment;
4. no excessive spasticity in any of the joints of the affected arm (shoulder, elbow, wrist, and fingers);
5. able to follow instructions and perform the study tasks (Mini Mental State Examination ≥ 22);
6. without upper extremity fracture within 3 months;
7. no participation in any rehabilitation experiments or drug studies during the study period; and (8) willing to provide written informed consent.

Exclusion Criteria:

1. acute inflammatory disease;
2. major health problems or poor physical condition that might limit participation; and (3) attend any other study in recent 3 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer assessment(FMA) | baseline, 3 weeks, 6 weeks, 18 weeks

SECONDARY OUTCOMES:
Wolf Motor Function Test (WMFT) | baseline, 6 weeks
Change scores of Box and block test (BBT) | baseline, 3 weeks, 6 weeks, 18 weeks
Change scores of Action research arm test (ARAT) | baseline, 3 weeks, 6 weeks
Change scores of Medical Research Council scale (MRC) | baseline, 3 weeks, 6 weeks
Change scores of Modified Ashworth scale (MAS) | baseline, 3 weeks, 6 weeks
Change scores of Myoton | baseline, 6 weeks
Change scores of Chedoke Arm and Hand Activity Inventory (CAHAI) | baseline, 6 weeks
Change scores of Functional independent measure (FIM) | baseline, 3 weeks, 6 weeks
Change scores of Stroke Impact Scale (SIS 3.0 version) | baseline, 3 weeks, 6 weeks, 18 weeks
Change scores of EuroQol Quality of Life Scale (EQ-5D) | baseline, 6 weeks
Change scores of Hand strength | baseline, 3 weeks, 6 weeks
Change scores of Motor activity log (MAL) | baseline, 6 weeks, 18 weeks
Change scores of ABILHAND Questionnaire | baseline, 6 weeks, 18 weeks
Change scores of 10-meter walking test | baseline, 6 weeks
Change scores of Nottingham Extended ADL Questionnaire (NEADL) | baseline, 6 weeks, 18 weeks
Change scores of Adelaide Activities Profile (AAP) | baseline, 6 weeks
Change scores of Accelerometer | baseline, 6 weeks
Change scores of kinematic analysis | baseline, 6 weeks
Change scores of Adverse effects | baseline, 3 weeks, 6 weeks
Change scores of Algometer | baseline, 6 weeks
Change scores of Revised Nottingham Sensory Assessment (rNSA) | baseline, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (3):
- Taiwan (3):
  - Lo-Sheng Sanatorium and Hospital, Kwei-shan, Toayuan County
  - Chang Gung Memorial Hospital, Kwei-Shan, Tao-Yuan
  - Taipei Hospital, Ministry of Health and Welfare, New Taipei City

REFERENCES:
- [Derived] Hung CS, Lin KC, Chang WY, Huang WC, Chang YJ, Chen CL, Grace Yao K, Lee YY. Unilateral vs Bilateral Hybrid Approaches for Upper Limb Rehabilitation in Chronic Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Dec;100(12):2225-2232. doi: 10.1016/j.apmr.2019.06.021. Epub 2019 Aug 14. PMID 31421096